CLINICAL TRIAL: NCT01000025
Title: A Double Blind Placebo Controlled Randomized Trial of PF-804 in Patients With Incurable Stage IIIB/IV Non-Small Cell Lung Cancer After Failure of Standard Therapy for Advanced or Metastatic Disease
Brief Title: PF-00299804 in Stage IIIB or Stage IV Non-Small Cell Lung Cancer Not Responding to Standard Therapy for Advanced or Metastatic Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: NCIC Clinical Trials Group (Network)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Organization: Canadian Cancer Trials Group (Network)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BR26; CAN-NCIC-BR26 (Other: PDQ); PFIZER-CAN-NCIC-BR26 (Other: Pfizer); CDR0000657246 (Other: PDQ)
Record Dates: First submitted 2009-10-21; First posted 2009-10-22 (Estimated); Results first posted 2014-10-27 (Estimated); Last update posted 2023-08-22 (Actual); Status verified 2020-04

CONDITIONS: Lung Cancer
Keywords: stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer; recurrent non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — dacomitinib

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- PF-00299804 (Active Comparator): Patients receive oral PF-00299804 once daily. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: PF-00299804
- Placebo (Placebo Comparator): Patients receive oral placebo once daily. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PF-00299804 — PF-804 45 mg PO, daily
  Arms: PF-00299804
Drug: Placebo — Placebo 45 mg PO, daily
  Arms: Placebo

SUMMARY:
RATIONALE: PF-00299804 may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. It is not yet known whether PF-00299804 is more effective than a placebo in treating patients with advanced non-small cell lung cancer.

PURPOSE: This randomized phase III trial is studying PF-00299804 to see how well it works compared with a placebo in treating patients with stage IIIB or stage IV non-small cell lung cancer that has not responded to standard therapy for advanced or metastatic cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To compare overall survival in patients with incurable stage III or IV non-small cell lung cancer receiving PF-00299804 versus placebo after failure of standard therapy for advanced metastatic disease.

Secondary

* To compare overall survival in KRAS-WT patients between the two arms.
* To compare overall survival in EGFR-mutant patients between the two arms.
* To compare progression-free survival between arms.
* To compare objective response rates between arms.
* To estimate time to response and response duration in these patients.
* To evaluate the nature, severity, and frequency of toxicities between arms.
* To compare quality of life between arms.
* To determine the incremental cost-effectiveness and cost-utility ratios for PF-00299804.
* To correlate the expression of tumor and blood markers (at diagnosis) with outcomes and response.

OUTLINE: This is a multicenter study. Patients are stratified according to center, performance status (0 or 1 vs 2 or 3), tobacco use (never vs past or present), best response to prior EGFR tyrosine kinase inhibitor (progressive disease vs other), weight loss (< 5% vs ≥ 5% or unknown), and ethnicity (East Asian vs other). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive oral PF-00299804 once daily. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity.
* Arm II: Patients receive oral placebo once daily. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity.

Blood, serum, plasma, and tissue samples are collected and examined for biomarkers and gene mutations, and may be banked for future studies.

Patients complete quality-of-life questionnaires EORTC QLQ-C30 and other questionnaires at baseline and then periodically during and after completion of study treatment.

Cost effectiveness and cost utility of PF-00299804 is assessed via the Health Utilities Index (EQ-5D) and the Resource Utilization Assessment periodically.

After completion of study treatment, patients are followed at 4 weeks and then every 12 weeks thereafter.

ELIGIBILITY:
Eligibility Criteria

* Histologically confirmed diagnosis of non-small cell carcinoma of the lung. Patients must have an adequate histopathology or cytology specimen must consent to release of all specimens for this protocol, and the centre/pathologist must have agreed to submission of the specimens.
* Patients must have evidence of disease, but measurable disease is not mandatory. To be considered evaluable for complete or partial response assessment, patients must have at least one measurable lesion as follows:

X-ray ≥ 20 mm Spiral CT scan or physical exam ≥ 10 mm (lymph nodes must be ≥ 15 mm in the short axis); Measurable lesions must be outside a previous radiotherapy field if they are the sole site of disease, unless disease progression has been documented.

* Male or female, 18 years of age or older.
* ECOG performance status of 0, 1, 2 or 3. Patients with performance status of 3 are eligible providing that the investigator attests that the patient has a reasonable life expectancy (≥ 6 weeks).
* Adequate renal and hepatic functions as defined by the following required laboratory values obtained within 14 days prior to randomization. If anemic, patients should be asymptomatic and should not be decompensated.

Creatinine <1.5 upper limit of normal Total bilirubin < 1.5 upper limit of normal ALT (SGPT) < 2.5 times the upper limit of normal. Note: If clearly attributable to liver metastasis, ALT (SGPT) values < 5 times the upper limit of normal are permitted.

- Previous Therapy Failure of a treatment regimen is defined as the inability to continue a regimen for any reason including, but not limited to, progressive disease, toxicity, or patient request. Up to a maximum of three lines of chemotherapy for advanced/metastatic disease (defined below) and at least one of erlotinib or gefitinib for advanced/ metastatic disease (defined below) should have failed.

Exchange of one chemotherapy agent for another within a combination chemotherapy regimen is not considered a new regimen in the following circumstances

* carboplatin is substituted for cisplatin due to nephrotoxicity
* one agent in the combination regimen is changed due to hypersensitivity occurring in the first cycle.

Chemotherapy for Advanced/Metastatic Disease:

Patients must have recovered from any reversible toxic effects and at least 21 days must have elapsed from the last dose and prior to randomization (14 days from the last dose for chemotherapy regimens administered on a weekly schedule). Further palliative cytotoxic chemotherapy must not be planned.

Patients < 70 years:

• Must have received 1 and up to a maximum of 3prior chemotherapy regimens (at least one of the three must have been a combination regimen and at least one must have contained platinum).

Patients ≥ 70 years (generally accepted as being at the time of the administration of the first regimen of chemotherapy for advanced disease):

• Must have received 1 and up to a maximum of 3 prior chemotherapy regimens for their disease. These may have been single agent chemotherapy regimens and a platinum agent is not required in keeping with current standards of practice.

Adjuvant Chemotherapy: Patients may ALSO have had prior adjuvant therapy for completely resected disease, providing completed at least 12 months prior to randomization. Adjuvant regimens < 12 months prior to randomization and combined chemotherapy/radiation regimens for irresectable locally advanced stage III disease (irrespective of timing), are considered to be for advanced/metastatic disease and constitute one of the 3 permissible regimens. Patients must have recovered from any reversible treatment related toxicities prior to randomization.

EGFR Inhibitor Therapy: Patients may only be enrolled after failure of prior gefitinib or erlotinib for advanced or metastatic disease. Patients who have received adjuvant gefitinib or erlotinib for completely resected NSCLC and who have recurred < 12 months after discontinuing erlotinib or gefitinib are eligible. Patients who received gefitinib or erlotinib for neoadjuvant therapy only are not eligible. EGFR inhibitor therapy must have been discontinued at least 21 days prior to randomization. Patients who discontinued prior gefitinib or erlotinib therapy for severe or life threatening organ toxicity are not eligible. Patients may also have received other EGFR active agents (such as reversible oral agents or monoclonal antibodies or vaccines) in addition to erlotinib or gefitinib but may not have received ANY prior irreversible EGFR inhibitor such as BIBW2992, HKI-272 (neratinib).

Maintenance Therapy: The same chemotherapy or agent/s continued for longer than 4-6 cycles for the purposes of 'maintenance' is considered one regimen; if another chemotherapy agent is given with 'maintenance' intent, it is considered a second regimen providing that 'failure' is documented. Patients who received erlotinib or gefitinib with 'maintenance' intent after completion of 1st line chemotherapy are eligible providing that 'failure' is documented.

Radiation: Patients may have had prior radiation therapy provided that a minimum of 14 days has elapsed between the end of radiotherapy and randomization onto the study. (Exceptions may be made however, for low dose, non-myelosuppressive radiotherapy. Patients must have recovered from any acute toxic effects from radiation prior to randomization.

Previous Surgery: Previous surgery is permitted provided that wound healing has occurred and at least 14 days have elapsed (major surgery).

* Patient able (i.e. sufficiently fluent) and willing to complete the quality of life questionnaires. The baseline assessment must already have been completed. Inability (illiteracy, loss of sight, or other equivalent reason) to complete the questionnaires will not make the patient ineligible for the study. However, ability but unwillingness to complete the questionnaires will make the patient ineligible.
* Patient consent must be appropriately obtained in accordance with applicable local and regulatory requirements. Each patient must sign a consent form prior to enrollment in the trial to document their willingness to participate.
* Patients must be accessible for treatment and follow-up. All randomized patients must be followed and treated at participating centres. Investigators must assure themselves the patients randomized on this trial will be available for complete documentation of the treatment, adverse events, and follow-up.
* In accordance with NCIC CTG policy, protocol treatment is to begin within 2 working days of patient randomization.

Ineligibility Criteria

Patients who fulfill any of the following criteria are not eligible for admission to the study:

* Patients receiving concurrent treatment with other experimental drugs or anti-cancer therapy.
* Patients who have experienced untreated and/or uncontrolled cardiovascular conditions and/or have symptomatic cardiac dysfunction (unstable angina, congestive heart failure, myocardial infarction within the previous year or cardiac ventricular arrhythmias requiring medication, history of 2nd or 3rd degree atrioventricular conduction defects). Patients with a significant cardiac history, even if controlled, should have a LVEF > 50%.
* Patients with untreated brain or meningeal metastases are not eligible (CT scans are not required to rule this out unless there is a clinical suspicion of CNS disease). Patients with treated CNS disease who have radiologic or clinical evidence of stable brain metastases, with no evidence of cavitation or hemorrhage in the brain lesion, are eligible providing that they are asymptomatic and do not require corticosteroids (must have discontinued steroids at least 1 week prior to randomization).
* Patients with active or uncontrolled infections, or with serious illnesses or medical conditions which would not permit the patient to be managed according to the protocol, including

  * Severe dry eye syndrome
  * Keratoconjunctivitis sicca
  * Sjogren's syndrome
  * Severe exposure keratopathy
  * Disorders that might increase the risk for epithelium-related complications (e.g., bullous keratopathy, aniridia, severe chemical burns, neutrophilic keratitis)
  * Uncontrolled inflammatory gastrointestinal diseases (Crohn's, ulcerative colitis etc.)
  * Prior pneumonitis/ILD secondary to EGFR inhibitors
* Mean QTc with Bazetts correction > 470msec in screening ECG or history of familial long QT syndrome.
* Drugs that are highly dependent on CYP2D6 for metabolism are prohibited, since PF-804 is a potent CYP2D6 inhibitor in in vitro assays. These inhibitors or inducers are prohibited from 7 days prior to the first dose until the end of treatment with PF-804. These include: S-metoprolol, propafenone, timolol, amitriptyline, clomipramine, desipramine, imipramine, paroxetine, haloperidol, risperidone, thioridazine, codeine, flecainide, mexilletine, tamoxifen, venlafaxine. Lidocaine may be used with clinical monitoring (including telemetry). Opiates such as morphine, oxycodone, dihydrocodeine, hydrocodone, and tramadol can be used as substitutes to replace codeine. Use of these opiates should be monitored for altered analgesia during treatment with PF-804 as they may be partly metabolized by CYP2D6. If PF-804 is administered with drugs which are P-glycoprotein (P-gp) substrates and have a narrow therapeutic index, monitoring for exaggerated effect and/or toxicities is recommended.
* Pregnancy or inadequate contraception. Women must be post-menopausal, surgically sterile, or use two reliable forms of contraception. Women of child-bearing potential must have a pregnancy test taken and proven negative within 7 days prior to randomization. Men must be surgically sterile or use a barrier method of contraception.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 720 (Actual)
Dates: Start 2009-12-23 (Actual); Primary Completion 2014-01-15 (Actual); Study Completion 2015-11-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Ellis, MD, Study Chair — Margaret and Charles Juravinski Cancer Centre; Penny Bradbury, MD, Study Chair — NCIC Clinical Trials Group; Michael Millward, MD, Study Chair — Sir Charles Gairdner Hospital - Nedlands
Locations (89):
- United States (2):
  - Shapiro, Stafford and Yee, Arcadia, California
  - Clintell, Inc., Skokie, Illinois
- Argentina (4):
  - CER - Instituto Medico, Buenos Aires, B1878dvb Bs. As.
  - COIBA Centro de Oncologia e Investigacion, Berazategui, Buenos Aires
  - Damic-Fundacion Rusculleda, Córdoba
  - Centro Medico San Roque, San Miguel de Tucumán
- Australia (16):
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - Concord Repatriation General Hospital, Concord, New South Wales
  - St. George Hospital, Cancer Care Centre, Kogarah, New South Wales
  - Prince of Wales Hospital, Randwick, New South Wales
  - Royal North Shore Hospital, St Leonards, New South Wales
  - Calvary Mater Newcastle Hospital, Waratah, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - The Prince Charles Hospital, Chermside, Queensland
  - Nambour General Hospital, Nambour, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Monash Medical Centre, Clayton, Victoria
  - Western Hospital, Footscray, Victoria
  - Frankston Hospital - Peninsula Oncology Centre, Frankston, Victoria
  - Geelong Hospital, Geelong, Victoria
  - Austin Hospital, Heidelberg, Victoria
  - Sir Charles Gairdner Hospital, Perth, Western Australia
- Brazil (8):
  - Centro de Oncologia e Radioterapia (COR) Mae de Deus, Porto Alegre, Rio Grande do Sul
  - Fundacao Pio XII - Hospital de Cancer de Barretos, Barretos, São Paulo
  - ESHO - Empresa de Servicos Hospitalares Ltda., Brasilia, São Paulo
  - Centro de Pesquisa Clinica do Hospital, Porto Alegre, São Paulo
  - Oxion Hospital Dia Oncologia LTDA - Oxion, Belo Horizonte
  - Centro
  - Nucleo de Oncologia da Bahia, Salvador
  - GRAM - Grupo de Assistencia Medica, São Paulo
- Canada (21):
  - Cross Cancer Institute, Edmonton, Alberta
  - BCCA - Abbotsford Centre, Abbotsford, British Columbia
  - BCCA - Fraser Valley Cancer Centre, Surrey, British Columbia
  - BCCA - Vancouver Cancer Centre, Vancouver, British Columbia
  - Atlantic Health Sciences Corporation, Saint John, New Brunswick
  - Dr. H. Bliss Murphy Cancer Centre, St. John's, Newfoundland and Labrador
  - QEII Health Sciences Centre, Halifax, Nova Scotia
  - Health Sciences North, Greater Sudbury, Ontario
  - Juravinski Cancer Centre at Hamilton Health Sciences, Hamilton, Ontario
  - Cancer Centre of Southeastern Ontario at Kingston, Kingston, Ontario
  - London Regional Cancer Program, London, Ontario
  - Lakeridge Health Oshawa, Oshawa, Ontario
  - Ottawa Health Research Institute - General Division, Ottawa, Ontario
  - Algoma District Cancer Program, Sault Ste. Marie, Ontario
  - Niagara Health System, St. Catharines, Ontario
  - Univ. Health Network-Princess Margaret Hospital, Toronto, Ontario
  - Windsor Regional Cancer Centre, Windsor, Ontario
  - CHUM - Hopital Notre-Dame, Montreal, Quebec
  - McGill University - Dept. Oncology, Montreal, Quebec
  - Allan Blair Cancer Centre, Regina, Saskatchewan
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan
- Italy (19):
  - Centro di Riferimento Oncologico - CRO, Aviano, PN
  - A.O. Busto Arsizio - P.O. Saronno, Saronno, VA
  - U.O. di Oncologia Medica Azienda Ospedaliera G Rummo, Benevento
  - Ospedale Santa Croce, Fano
  - U.O. di Oncologia Ospedale Villa Scassi, Genova
  - Intstituto Scientifico Romangnolo, Meldola
  - U.O.C. Terapie Integrate in Oncologia,, Messina
  - U.O.C. Oncologia Medica,, Messina
  - Ospedale San Raffaele, Milan
  - U.O.C. di Oncologia U.L.S.S. 13, Mirano
  - Dott. Fortunato Ciardiello,Cattedra Oncologia Medica, Napoli
  - Unita Sperimentazioni Cliniche Istituto per lo, Napoli
  - UOC Oncologia Medica II Instituto Oncologio Veneto, Padua
  - La Maddalena, Dipartimento Oncologico, Palermo
  - Azienda USL di Piacenza, Ospedale Gugliemimo Salieto, Piacenza
  - Azienda Ospedaliera S. Camillo-Forlanin, Rome
  - Policlinico Umberto I, Universita Sapienza, Rome
  - Ospedale Casa Sollievo della Sofferenza, San Giovanni Rotondo
  - Ospedale E. Morelli-Sondalo, Sondalo
- Auckland City Hospital, Auckland, New Zealand
- Peru (3):
  - Hospital Central De La Fuerza Aerea Del Peru, Lima
  - Hospital Nacional Luis N. Saenz, Lima
  - Instituto de Oncologia y Radioterapia de, Lima
- Philippines (3):
  - Perpetual Succour Hospital, Cebu City
  - Makati Medical Center, Makati City
  - Phillippine General Hospital, Manila
- South Korea (5):
  - Ajou University Hospital, Gyeonggi-do
  - Chonnan National University Hwasun Hospital, Jeongnam
  - Yonsei University College of Medicine, Seoul
  - Seoul Veterans Hospital, Seoul
  - The Catholic University of Korea,, Seoul
- Taiwan (3):
  - China Medical University Hospital, Taichung
  - Chi-Mei Foundation Hospital, Tainan
  - Tri-Service General Hospital, Taipei
- Thailand (4):
  - Chulalongkorn University, Bangkok
  - Ramathibodi Hospital, Bangkok
  - Siriraj Hospital, Oncology Unit, Bangkok
  - Maharaj Nakorn Chiangmai Hospital, Chiang Mai

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ellis PM, Shepherd FA, Millward M, Perrone F, Seymour L, Liu G, Sun S, Cho BC, Morabito A, Leighl NB, Stockler MR, Lee CW, Wierzbicki R, Cohen V, Blais N, Sangha RS, Favaretto AG, Kang JH, Tsao MS, Wilson CF, Goldberg Z, Ding K, Goss GD, Bradbury PA; NCIC CTG; Australasian Lung Cancer Trials Group; NCI Naples Clinical Trials Unit. Dacomitinib compared with placebo in pretreated patients with advanced or metastatic non-small-cell lung cancer (NCIC CTG BR.26): a double-blind, randomised, phase 3 trial. Lancet Oncol. 2014 Nov;15(12):1379-88. doi: 10.1016/S1470-2045(14)70472-3. Epub 2014 Oct 15. PMID 25439692
- [Derived] Martin P, Shiau CJ, Pasic M, Tsao M, Kamel-Reid S, Lin S, Tudor R, Cheng S, Higgins B, Burkes R, Ng M, Arif S, Ellis PM, Hubay S, Kuruvilla S, Laurie SA, Li J, Hwang D, Lau A, Shepherd FA, Le LW, Leighl NB. Clinical impact of mutation fraction in epidermal growth factor receptor mutation positive NSCLC patients. Br J Cancer. 2016 Mar 15;114(6):616-22. doi: 10.1038/bjc.2016.22. Epub 2016 Feb 18. PMID 26889973

RESULTS

PARTICIPANT FLOW:
Groups:
- PF-804: Study treatment arm
- Placebo: Control arm
Period: Overall Study
Arm/Group | PF-804 | Placebo
Started | 480 | 240
Completed | 12 | 2
Not Completed | 468 | 238
Not completed — Adverse Event | 43 | 2
Not completed — Withdrawal by Subject | 13 | 8
Not completed — Death | 23 | 13
Not completed — Lack of Efficacy | 363 | 208
Not completed — Intercurrent Illness | 26 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PF-00299804 | Placebo | Total
Number analyzed (Participants) | 480 | 240 | 720
Age, Continuous [Median (Full Range); unit: years] | 63.5 [32 to 86] | 65.5 [34 to 90] | 64 [32 to 90]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 236 | 120 | 356
  Male | 244 | 120 | 364
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 2
  Asian | 172 | 87 | 259
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 4 | 1 | 5
  White | 288 | 144 | 432
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 13 | 8 | 21
Region of Enrollment [Number; unit: participants]
  United States | 1 | 1 | 2
  Philippines | 20 | 11 | 31
  Taiwan | 11 | 6 | 17
  Canada | 207 | 101 | 308
  Thailand | 28 | 14 | 42
  Brazil | 25 | 14 | 39
  Peru | 0 | 1 | 1
  Australia | 50 | 27 | 77
  New Zealand | 7 | 4 | 11
  Italy | 77 | 34 | 111
  Korea, Republic of | 47 | 24 | 71
  Argentina | 7 | 3 | 10

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: Median and 95% confidence intervals
Time Frame: 42 Months
Population: ITT
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | PF-00299804 | Placebo
Number analyzed (Participants) | 480 | 240
Months | 6.83 [6.08 to 7.49] | 6.31 [5.32 to 7.52]
Statistical Analysis 1: Comparison: PF-00299804 vs Placebo; The trial was designed to detect a 25% deduction in risk of death with PF-804 with 90% power using a 1-sided 2.5% level significance test. The sample size was estimated as 720 patients; Test type: Superiority or Other; p = 0.506, Log Rank — Stratified by stratification factors at randomization except study center, but included K-Ras mutation status.1-sied p-value; Stratified by stratification factors at randomization except study center, but included K-Ras mutation status; Hazard Ratio (HR) = 1.00, 95% CI 2-sided [0.83 to 1.21]

2. Secondary Outcome: Overall Survival in KRAS-WT Patients
Description: Median and 95% confidence intervals of Overall survival in KRAS-WT patients
Time Frame: 42 Months
Population: Patients with K-Ras mutation wild type
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | PF-00299804 | Placebo
Number analyzed (Participants) | 220 | 120
Months | 7.00 [6.01 to 8.21] | 5.19 [4.53 to 7.00]
Statistical Analysis 1: Comparison: PF-00299804 vs Placebo; Test type: Superiority or Other; p = 0.043, Log Rank — 1-sided p-value; Stratified by stratification factors at randomization except study center; Hazard Ratio (HR) = 0.79, 95% CI 2-sided [0.61 to 1.03]

3. Secondary Outcome: Overall Survival in EGFR-mutant Patients
Description: Overall survival by EGFR-mutantion subgroups
Time Frame: 42 Months
Population: Patients with EGFR mutation
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | PF-00299804 | Placebo
Number analyzed (Participants) | 114 | 68
Months | 7.23 [6.08 to 8.61] | 7.52 [4.99 to 9.49]
Statistical Analysis 1: Comparison: PF-00299804 vs Placebo; Test type: Superiority or Other; p = 0.46, Log Rank — 1-sided pvalue; Hazard Ratio (HR) = 0.98, 95% CI 2-sided [0.67 to 1.44]

4. Secondary Outcome: Progression-free Survival
Description: progression were evaluated using the revised international criteria (1.1) proposed by the RECIST (Response Evaluation Criteria in Solid Tumours) committee
Time Frame: 42 Months
Population: ITT
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | PF-00299804 | Placebo
Number analyzed (Participants) | 480 | 240
Months | 2.66 [1.91 to 3.32] | 1.58 [0.99 to 1.74]
Statistical Analysis 1: Comparison: PF-00299804 vs Placebo; Test type: Superiority or Other; p < 0.0001, Log Rank; Stratified by stratification factors at randomization except study center, but included K-Ras mutation status; Hazard Ratio (HR) = 0.66, 95% CI 2-sided [0.55 to 0.79]

5. Secondary Outcome: Objective Response Rate
Description: Response were evaluated in this study using the revised international criteria (1.1) proposed by the RECIST (Response Evaluation Criteria in Solid Tumours) committee. BEST RESPONSE from the start of study treatment until the end of treatment were reported.Objective response rate is the sum of CR + PR divided by the total number of patients in each group.
Time Frame: 42 months
Population: ITT
Measure: Mean (95% Confidence Interval); unit: percentage of participants
Arm/Group | PF-00299804 | Placebo
Number analyzed (Participants) | 480 | 240
percentage of participants | 7.1 [4.8 to 9.4] | 1.3 [0.0 to 2.7]
Statistical Analysis 1: Comparison: PF-00299804 vs Placebo; Test type: Superiority or Other; p = 0.001, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 6.11, 95% CI 2-sided [1.84 to 20.3]

6. Secondary Outcome: Number of Participants With Toxicity as Measured by NCI CTCAE Version 4.0
Description: Number of participants with Toxicities by treatment received according to NCI CTCAE version 4.0
Time Frame: 42 Months
Population: As treated population
Measure: Number; unit: participants
Arm/Group | PF-00299804 | Placebo
Number analyzed (Participants) | 477 | 239
participants | 467 | 223

ADVERSE EVENTS:
Time Frame: 42 Months
Arm/Group | PF-00299804 | Placebo
Serious Adverse Events (participants affected / at risk) | 191/477 | 87/239
Other Adverse Events (participants affected / at risk) | 465/477 | 219/239
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PF-00299804 (N=477) | Placebo (N=239)
Anemia (Blood and lymphatic system disorders) | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 1
Pericardial effusion (Cardiac disorders) | 1 | 2
Pericardial tamponade (Cardiac disorders) | 0 | 1
Pericarditis (Cardiac disorders) | 1 | 0
Hearing impaired (Ear and labyrinth disorders) | 1 | 0
Adrenal insufficiency (Endocrine disorders) | 0 | 1
Cataract (Eye disorders) | 1 | 0
Corneal ulcer (Eye disorders) | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 4 | 3
Anal hemorrhage (Gastrointestinal disorders) | 1 | 0
Ascites (Gastrointestinal disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 1 | 0
Colonic obstruction (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 3 | 0
Diarrhea (Gastrointestinal disorders) | 17 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 2
Esophageal stenosis (Gastrointestinal disorders) | 0 | 1
Gastrointestinal pain (Gastrointestinal disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 0 | 1
Mucositis oral (Gastrointestinal disorders) | 5 | 0
Nausea (Gastrointestinal disorders) | 5 | 0
Obstruction gastric (Gastrointestinal disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 8 | 3
Chills (General disorders) | 1 | 0
Death NOS (General disorders) | 2 | 0
Fatigue (General disorders) | 4 | 2
Fever (General disorders) | 7 | 1
Gait disturbance (General disorders) | 1 | 0
Infusion site extravasation (General disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 1 | 0
Pain (General disorders) | 2 | 1
Sudden death NOS (General disorders) | 1 | 2
Hepatic failure (Hepatobiliary disorders) | 1 | 0
Bronchial infection (Infections and infestations) | 1 | 1
Enterocolitis infectious (Infections and infestations) | 1 | 0
Lung infection (Infections and infestations) | 32 | 12
Lymph gland infection (Infections and infestations) | 1 | 0
Mucosal infection (Infections and infestations) | 1 | 0
Other infections and infestations (Infections and infestations) | 1 | 0
Scrotal infection (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 2 | 3
Skin infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 2 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0
Fracture (Injury, poisoning and procedural complications) | 3 | 1
Hip fracture (Injury, poisoning and procedural complications) | 3 | 0
Neutrophil count decreased (Investigations) | 0 | 1
Weight loss (Investigations) | 0 | 1
Anorexia (Metabolism and nutrition disorders) | 3 | 1
Dehydration (Metabolism and nutrition disorders) | 16 | 0
Hypercalcemia (Metabolism and nutrition disorders) | 0 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatremia (Metabolism and nutrition disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 0
Other neoplasms benign, malignant and unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 79 | 43
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Cognitive disturbance (Nervous system disorders) | 0 | 1
Depressed level of consciousness (Nervous system disorders) | 4 | 0
Dizziness (Nervous system disorders) | 2 | 1
Dysphasia (Nervous system disorders) | 1 | 0
Encephalopathy (Nervous system disorders) | 1 | 0
Intracranial hemorrhage (Nervous system disorders) | 0 | 1
Ischemia cerebrovascular (Nervous system disorders) | 1 | 0
Other nervous system disorders (Nervous system disorders) | 1 | 0
Paresthesia (Nervous system disorders) | 0 | 1
Seizure (Nervous system disorders) | 1 | 0
Sinus pain (Nervous system disorders) | 1 | 0
Stroke (Nervous system disorders) | 2 | 3
Syncope (Nervous system disorders) | 0 | 1
Transient ischemic attacks (Nervous system disorders) | 0 | 1
Confusion (Psychiatric disorders) | 3 | 1
Personality change (Psychiatric disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 6 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 6 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 26 | 14
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 7 | 3
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 6 | 2
Other skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 2 | 1
Rash acneiform (Skin and subcutaneous tissue disorders) | 2 | 0
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 1 | 0
Hypotension (Vascular disorders) | 0 | 1
Other vascular disorders (Vascular disorders) | 0 | 1
Thromboembolic event (Vascular disorders) | 12 | 3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PF-00299804 (N=477) | Placebo (N=239)
Conjunctivitis (Eye disorders) | 47 | 0
Dry eye (Eye disorders) | 41 | 5
Abdominal pain (Gastrointestinal disorders) | 61 | 18
Constipation (Gastrointestinal disorders) | 120 | 74
Diarrhea (Gastrointestinal disorders) | 380 | 47
Dry mouth (Gastrointestinal disorders) | 50 | 11
Dyspepsia (Gastrointestinal disorders) | 39 | 12
Gastroesophageal reflux disease (Gastrointestinal disorders) | 30 | 9
Mucositis oral (Gastrointestinal disorders) | 206 | 8
Nausea (Gastrointestinal disorders) | 168 | 59
Vomiting (Gastrointestinal disorders) | 134 | 37
Edema limbs (General disorders) | 57 | 28
Fatigue (General disorders) | 254 | 115
Fever (General disorders) | 42 | 15
Non-cardiac chest pain (General disorders) | 33 | 21
Pain (General disorders) | 93 | 50
Lung infection (Infections and infestations) | 25 | 6
Paronychia (Infections and infestations) | 142 | 0
Weight loss (Investigations) | 73 | 23
Anorexia (Metabolism and nutrition disorders) | 222 | 93
Back pain (Musculoskeletal and connective tissue disorders) | 83 | 47
Bone pain (Musculoskeletal and connective tissue disorders) | 48 | 20
Chest wall pain (Musculoskeletal and connective tissue disorders) | 41 | 27
Pain in extremity (Musculoskeletal and connective tissue disorders) | 79 | 35
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 31 | 13
Dizziness (Nervous system disorders) | 55 | 25
Dysgeusia (Nervous system disorders) | 34 | 4
Headache (Nervous system disorders) | 53 | 29
Peripheral sensory neuropathy (Nervous system disorders) | 84 | 32
Anxiety (Psychiatric disorders) | 30 | 20
Insomnia (Psychiatric disorders) | 84 | 45
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 25 | 14
Cough (Respiratory, thoracic and mediastinal disorders) | 233 | 108
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 276 | 132
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 72 | 4
Productive cough (Respiratory, thoracic and mediastinal disorders) | 58 | 32
Sore throat (Respiratory, thoracic and mediastinal disorders) | 26 | 3
Alopecia (Skin and subcutaneous tissue disorders) | 25 | 11
Dry skin (Skin and subcutaneous tissue disorders) | 171 | 27
Other skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 30 | 5
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 55 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 87 | 28
Rash acneiform (Skin and subcutaneous tissue disorders) | 283 | 24
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 78 | 16

LIMITATIONS AND CAVEATS:
Despite the eligibility requirement for tumor samples, samples were not available or inadequate for translational studies in 30 - 40% of patients. This does limits the power of the secondary analyses examining biomarker driven outcomes.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No